CLINICAL TRIAL: NCT03817541
Title: Expiratory and Plasma Propofol Concentration in Bariatric and Cholecystectomy Patients
Brief Title: Expiratory and Plasma Propofol Concentration in Gastrological Surgery Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Johan C Ræder, Professor, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Expiratory propofol gastro
Record Dates: First submitted 2019-01-18; First posted 2019-01-25 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Bariatric Surgery Candidate; Cholecystectomy

STUDY DESIGN:
Intervention Model Description: One Group of morbidly obese patients for bariatric surgery One Group of normal weight cholecystectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bariatric surgery (Experimental): Patients due for bariatric surgery, BMI > 30
  Interventions: Device: Edmon (reg), BBraun
- Cholecystectomy (Experimental): Normal weight patients due for cholecystectomies
  Interventions: Device: Edmon (reg), BBraun

INTERVENTIONS:
Device: Edmon (reg), BBraun — exhaled propofol will be compared With plasma propofol values
  Other Names: propofol plasma sample

SUMMARY:
Determination of accuracy With Edmond (reg) expiratory propofol measurement Device, compared With concommitant plasma samples of propofol

DETAILED DESCRIPTION:
Edmon (trade mark) is a New Device from BBraun, measuring the expiratory concentration of propofol in anaesthetized patients.

The investigators will test the accuracy and stability of such measurements in comparison With plasma propofol Levels.

The investigators will test during target Control infusion (Marsh model) and assumed stable plasma Levels.

Plasma samples of propofol will be taken for comparison With exhaled propofol.

ELIGIBILITY:
Inclusion Criteria:

* • Patients admitted to Oslo University Hospital, scheduled for elective laparoscopic bariatric surgery or elective laparoscopic cholecystectomy.

  * Both genders.
  * Age 18-60 years, both inclusive.
  * BMI ≥ 20 kg/m2, 10 patients with BMI 20-30, and 10 patients with BMI > 40
  * ASA classification I-III

Exclusion Criteria:

* • Known hypersensitivity or other contraindication to propofol administered as Target Controlled Infusion.

  * Patients which during a preoperative visit are deemed not to tolerate propofol bolus or infusion as administered by Target Controlled Infusion.
  * Ongoing neuroleptic medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
exhaled propofol concentration | start of anaesthesia to end of anaesthesia, 2-3 hours in total
  parts per billion
propofol plasma concentration | 4-6 samples in the period between start and end of anaesthesia
  microg pr ml

SECONDARY OUTCOMES:
calculated plasma concentration | From start of anaesthesia until end of anaesthesia, 1-3 hrs in total
  Marsh model prediction, microg pr ml
BIS | from start of anaesthesia until end of anaestheisa, 1-3 hours in total
  Bispectral index value, score = 0-100
calculated effect site concentration | from start of anaesthesia until end of anaesthesia, 1-3 hours in total
  Marsh model, microg pr ml
EEG Power spectrum | f
  Spectral edge value (Hz)
EEG Power distribution | from start of anaesthesia until end of anaesthesia, 1-3 hours in total
  % representation relative Power of Alpha, Beta, Theta, Gamma band

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Anesthesiology, Oslo University Hospital, Ullevaal, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided